CLINICAL TRIAL: NCT05883657
Title: Evaluation of the Tolerance and Performance of Cyto-selective Difluoroethane-based Cryotherapy in the Treatment of Brown Spots (Solar and Senile Lentigines, Post-Inflammatory Hyperpigmentation)
Brief Title: Tolerance and Performance of Cyto-selective Difluoroethane-based Cryotherapy in the Treatment of Brown Spots (Solar and Senile Lentigines, Post-Inflammatory Hyperpigmentation)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cryonove Pharma (Industry)
Collaborators: Dermatech (Industry); CEISO (Industry); Sefako Makgatho Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CS5_7
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-04

CONDITIONS: Solar Lentigo; Senile Lentigo; Post Inflammatory Hyperpigmentation
Keywords: Cryotherapy; Skin Disease; Hyperpigmentation
MeSH Terms: conditions — Hyperpigmentation; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Condition 1 : Prototypes (816-v1) every weeks (Experimental): Application on the brown spots of the face and the hands for the prototypes (816-v1) at D0, D7, D14, D21, D28, D35, D42, D49, D56, D63, D70 and D77.
  Interventions: Device: Condition 1 : Prototypes (816-v1) every weeks
- Condition 2 : Prototypes (816-v1) every two weeks (Experimental): Application on the brown spots of the face and the hands for the prototypes (816-v1) at D0, D14, D28, D42, D56 and D70.
  Interventions: Device: Condition 2 : Prototypes (816-v1) every two weeks

INTERVENTIONS:
Device: Condition 1 : Prototypes (816-v1) every weeks — Application on brown spots located on the face and/or the hand (12 treatments during the study). An operator previously trained by the dermatologist will apply the study device to the patient's face or/and hand. Subjects will be lying down, and the prototypes will be administered upside down for the applications on the face and sitting for the applications on the hands. For the application on the hands, the hands will be placed flat on the table and the prototypes will be applied upside down. During applications on the face, subjects will wear diving goggles protecting the eyes from cryogenic gas.
  Arms: Condition 1 : Prototypes (816-v1) every weeks
Device: Condition 2 : Prototypes (816-v1) every two weeks — Application on brown spots located on the face and/or the hand (6 treatments during the study). An operator previously trained by the dermatologist will apply the study device to the patient's face or/and hand. Subjects will be lying down, and the prototypes will be administered upside down for the applications on the face and sitting for the applications on the hands. For the application on the hands, the hands will be placed flat on the table and the prototypes will be applied upside down. During applications on the face, subjects will wear diving goggles protecting the eyes from cryogenic gas.
  Arms: Condition 2 : Prototypes (816-v1) every two weeks

SUMMARY:
CS5_7 study aim to evaluate the tolerance and to adjust the mode of administration of two conditions of cryotherapy treatment applied on the brown spots of the face and hands with 1 prototype (816-v1). A brown spot is defined as solar or senile lentigo and post-inflammatory hyperpigmentation (PIH).

The study will evaluate the following prototype :

• Prototypes from (816-v1 201) to (816-v1 290)

DETAILED DESCRIPTION:
Rational :

Hyperpigmentation is a problem in all skin types. Safe depigmentation is a challenge. Cryotherapy with liquid nitrogen at -70 °C has been used in the treatment of solar skin lesions for many years but causes considerable damage.

Solar/senile lentigo is a harmless patch of darkened skin. It results from exposure to ultraviolet (UV) radiation, which causes local proliferation of melanocytes and accumulation of melanin within the skin cells (keratinocytes). Solar/senile lentigos or lentigines are very common, especially in people over the age of 40 years.

A solar/senile lentigo is a flat, well-circumscribed patch. It can be round, oval or irregular in shape. Colour varies from skin-coloured, tan to dark brown or black, and size varies from a few millimetres to several centimetres in diameter. They can be slightly scaly. Solar/senile lentigines are found as groups of similar lesions on sun-exposed sites, particularly the face or the back of hands.

Cryotherapy is more and more used to improve skin appearance and currently used to treat lentigo spot. However, the cryogenic gas (conventional cryotherapy - liquid nitrogen) creates a dermabrasion of the skin surface and person receiving this kind of treatment presents an impaired skin during a few days following the treatment as temporary damage of stratum corneum, erythema, scars, burns

Following the side effects occurring after conventional cryotherapy application, the Sponsor has developed some devices using difluoroethane, manufactured by CRYONOVE PHARMA, already available on the local and international markets, e.g. CRYOBEAUTY MAINS and CRYOBEAUTY CORPS.

To continue its research and development activities, the sponsor has selected a new sequence of a specific cryogenic spray which has been used effectively and safely for lentigos treatment in Fitzpatrick phototypes I to IV on the face, with benefit for the subjects without any adverse safety outcomes. There is therefore a need to test the devices for lentigo and PIH on darker skin phototypes (V and VI according to Fitzpatrick scale), which also encounter hyperpigmentation challenges.

In the study, the clinical evaluation of different criteria performed by a Dermatologist before and after treatment will lead to objectively assess the safety (outcomes) and efficacy (depigmenting) of concerned criteria.

Design:

The study performed is a proof of performance designed to be interventional, monocentric, randomized and double blinded.

Intervention :

1 prototype of devices is evaluated in 2 conditions. Each treatment corresponds to a combination of a specific sequence of a cryogenic spray and of a frequency of application

At least 80 spots will be randomized between the 2 conditions. Prototypes (816-v1 201) to (816-v1 290) will be applied on brown spots located on the face and/or the hands .

In condition 1, each spots will be treated 12 times by a defined prototype (always the same device on the same spot all along the study) and according to specific frequencies (every week).

In condition 2, each spots will be treated 6 times by a defined prototype (always the same device on the same spot all along the study) and according to specific frequencies (every two weeks).

Prior to any study device application, the dermatologist will assess the adverse events and will decide if the period between two consecutive applications should be extended or not.The dermatologist will verify that the skin has not been treated by cosmetic products (no presence of cream that could interfere with the treatment) and is dry.

As the study will use prototypes, before each treatment, the prototype will be administered to any surface (in order to purge eventually the presence of air). An operator previously trained by the dermatologist will apply the study device to the patient's face.

Subjects will be lying down, and the device will be administered upside down. During applications on the face, subjects will wear diving goggles protecting the eyes from cryogenic gas. For the application on the hands, the hands will be placed flat on the table and the prototypes will be applied upside down.

The patient follow-up visits are from Day 0 to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Female or male.
* Ages 18 to 75.
* Phototypes V and VI (according with Fitzpatrick scale), according to the spots' distribution table.
* Featuring brown spots ≥ 3 and ≤ 6 mm in diameter (on the face (and when possible, on the hands).
* Agreeing not to be exposed to the sun (or artificial UV) during the study.
* Informed, having undergone a general clinical examination attesting to his/her ability to participate in the study.
* Having given written consent for their participation in the study.
* No suspicion of carcinoma after investigation by a dermatologist.

Exclusion Criteria:

* Having performed cosmetic treatments (exfoliants, scrubs or self-tanners, manicures (only nails care acceptable), facials, UV ...) in the month before the start of the study, at the level of the face and/or hands.
* Having applied a depilatoring product in the month prior to the start of the study, on the face and/or hands.
* Having performed cosmetic treatments in a dermatologist (laser, Intense Pulsed Light (IPL), peeling, creams, cryotherapy ...), on the face and/or hands in the last 6 months.
* With dermatosis, autoimmune disease, systemic, chronic or acute disease, or any other pathology that may interfere with treatment or influence the results of the study (people with diabetes or circulatory problems, allergic to cold, Raynaud's syndrome...).
* Receiving treatment by general or local (dermo corticoids, corticosteroids, diuretics ...) likely to interfere with the evaluation of the parameter studied.
* Participating in another study or being on a period of exclusion from a previous study.
* Unable to follow the requirements of the protocol.
* Vulnerable: whose ability or freedom to give or refuse consent is limited.
* Major protected by law (tutorship, curatorship, safeguarding justice...).
* People unable to read and write english language.
* Unable to be contacted urgently over the phone.

For female subjects:

* Pregnant woman (or wishing to be pregnant during study) or while breastfeeding.
* A woman who does not have a contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-10 (Estimated); Primary Completion 2023-12-12 (Estimated); Study Completion 2023-12-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline skin hyperpigmentation | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 63, Day 70, Day 77, Day 84 and Day 0 + 6 months
  The evaluation will be performed visually on the selected spots.
  A scale in 6 points (0 to 5) will be used :
  0=Clear of hyperpigmentation;
  1. Almost clear of hyperpigmentation;
  2. mild, but noticeable hyperpigmentation;
  3. moderate hyperpigmentation (medium brown in quality);
  4. severe hyperpigmentation (dark brown in quality);
  5. very severe hyperpigmentation (very dark brown, almost black in quality).
Change from baseline skin hypopigmentation | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 63, Day 70, Day 77, Day 84 and Day 0 + 6 months
  The evaluation will be performed visually on the selected spots.
  A scale in 5 points will be used (0 to 4):
  0=no hypopigmented lesion;
  1. very slight area of hypopigmentation of very small size and very slightly fairer than the surrounding skin;
  2. slight area of hypopigmentation of small size and slightly fairer than the surrounding skin;
  3. moderate : area of hypopigmentation of moderate size and much fairer than the surrounding skin;
  4. severe : area of hypopigmentation of large size and much fairer than the surrounding skin.
Change from baseline skin appearance | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 63, Day 70, Day 77, Day 84 and Day 0 + 6 months
  The evaluation will be performed visually on the selected spots and surrounded spotless skin area around the spot skin to assess erythema, oedema blister, bubble, scars, micro-bruise, hematoma, dryness,desquamation, fissures/cracks, roughness,crust, pink spots and papules.
  A scale in 5 points (0 to 4) will be used :
  0=none;
  1. very mild;
  2. mild;
  3. moderate;
  4. severe.
Change from baseline skin sensation | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 63, Day 70, Day 77, Day 84 and Day 0 + 6 months
  The evaluation will be performed visually on the selected spots and around the spot skin to assess tightness, stinging, itching, warm and burning sensation.
  A scale in 5 points (0 to 4) will be used :
  0=none;
  1. very mild;
  2. mild;
  3. moderate;
  4. severe.
Self-assesment of pain by VAS | Day 0
  The pain of the treatment will be assessed by the Visual Analogue Scale (VAS) at time T0 on the treated area.
  The pain assessed is that felt during the application of the devices. It will be collected from the patient within 5 minutes of application.
  The VAS is made up of a 10-centimeter line anchored by two ends of the pain. 10 is the first end being the "maximum pain imaginable" and 0 is the other end being "no pain".
Change from baseline spots visibility | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 63, Day 70, Day 77, Day 84 and Day 0 + 6 months
  Standardized photographs will be taken using a Dermatoscope C-Cube® (PIXIENCE) which allows realizing high resolution skin pictures. The capture will be taken on the previously selected lentigo and a spotless area.
Incidence of unexpected events | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 63, Day 70, Day 77, Day 84 and Day 0 + 6 months
  Unexpected events

SECONDARY OUTCOMES:
Self assessment of skin appearance | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 70, Day 84 and Day 0 + 6 months
  The skin appearance will be assessed by subjects through a 3 items questionnaire.
  It allows obtaining the subjective appraisal of subject on the treatments using the following 5-point scale:
  * agree,
  * quite agree
  * neither agree, nor disagree
  * quite disagree
  * disagree.
  The items are the following:
  * The spot seems clearer.
  * The size of the spot seems reduced.
  * The spot seems less visible.

CONTACTS AND LOCATIONS:
Overall Officials: Beverley Summers, Pr, Principal Investigator — Photobiology Laboratory
Locations (1):
- Photobiology Laboratory, Sefako Makgatho Health Sciences University, Pretoria, Gauteng, South Africa